CLINICAL TRIAL: NCT04821921
Title: The Impact of the COVID-19 Pandemic on Diabetes Management (CoDiaM)
Brief Title: The Impact of the COVID-19 Pandemic on Diabetes Management
Acronym: CoDiaM
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Dr. phil. Ingmar Schäfer, Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: IPA-2021-01
Record Dates: First submitted 2021-03-29; First posted 2021-03-30 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Type 2 Diabetes; Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with diabetes mellitus: Approximately 750 patients with diabetes mellitus from 3 GP practices specialized on diabetes treatment
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Care as usual

SUMMARY:
The "CoDiaM study" examines how diabetes management and outcomes are changing during the COVID-19 pandemic and whether these changes are influenced by socio-demographic factors, health literacy, self-efficacy and perceived social support.

DETAILED DESCRIPTION:
The Covid-19 pandemic created new challenges for patients with diabetes and their treating physicians. In order to protect people from SARS-COV-2 infections, social contacts were reduced by restrictions on many areas of social life. As a side effect, these measures could have also led to changes in the self-management of patients with diabetes mellitus, such as lack of physical exercise, less healthy dietary behavior, and a reduced intensity of medical care. These possible changes may be associated with poorer control of blood glucose, cholesterol, and blood pressure. Therefore, the CoDiaM study will investigate how management and outcomes of diabetes are changing during the pandemic and identify associated factors.

The study is based on data of patients treated in three GP practices specialized on diabetes treatment in Hamburg, Germany. Data collection will include a written patient survey and extraction of clinical data from patient records. The patient's survey includes sociodemographic data and validated instruments to assess diabetes self-management (DSMQ), health literacy (HLS-EU-Q16), self-efficacy (General Self-efficacy scale) and perceived social support (F-SozU K14). Data will be analyzed by descriptive statistics and multivariable, multilevel linear and logistic regression analyses adjusted for possible confounders and random effects on the practice level.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years or older, and
* having diabetes type 2 or type 1, and
* having consulted the practice at least once in 2019 AND at least once in 2020

Exclusion Criteria:

* no capacity to consent (e.g. because of dementia)
* insufficient German language skills to understand the questions in the questionnaire
* not able to fill out the questionnaire (e.g. because of blindness)
* gestational diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is located in Hamburg, Germany. Patients from three GP practices specialized on diabetes treatment in Hamburg will be included. In each practice, eligible patients with diabetes type 1 and 2 will receive patient information, consent form and questionnaire by mail. After written informed consent and after the questionnaires have been returned, data from patient records in the practices will be extracted. The investigators estimated that approximately 3000 patients will be eligible to be contacted. From pretest and experience with similar studies the investigators anticipated a response rate of 25% (=750 patients).
Sampling Method: Probability Sample
Enrollment: 1503 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c (HbA1c) | 01.01.2019 to 31.12.2021
  Data on outcome will be extracted from the GP's patient record

CONTACTS AND LOCATIONS:
Overall Officials: Ingmar Schäfer, Dr. phil., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Department of Primary Medical Care, University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No
Individual participant data are available from the principal investigator on reasonable request.

REFERENCES:
- [Derived] Tajdar D, Luhmann D, Walther L, Bittner L, Scherer M, Schafer I. Effects of Two COVID-19 Lockdowns on HbA1c Levels in Patients with Type 1 Diabetes and Associations with Digital Treatment, Health Literacy, and Diabetes Self-Management: A Multicenter, Observational Cohort Study Over 3 Years. Diabetes Ther. 2024 Jun;15(6):1375-1388. doi: 10.1007/s13300-024-01574-x. Epub 2024 Apr 20. PMID 38642263
- [Derived] Schafer I, Tajdar D, Walther L, Bittner L, Luhmann D, Scherer M. Impact of two COVID-19 lockdowns on HbA1c levels in patients with type 2 diabetes and associations with patient characteristics: a multicentre, observational cohort study over three years. Front Public Health. 2024 Jan 5;11:1272769. doi: 10.3389/fpubh.2023.1272769. eCollection 2023. PMID 38249413